CLINICAL TRIAL: NCT03861923
Title: Effectiveness of Dry Needling on Pain and Function for the Management of Shoulder Adhesive Capsulitis: a Randomized Controlled Trial
Brief Title: Dry Needling for Shoulder Adhesive Capsulitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00101726
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Shoulder Adhesive Capsulitis; Shoulder Pain; Frozen Shoulder
Keywords: dry needling; physical therapy; trigger point
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Dry Needling; Exercise Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling and exercise (Experimental)
  Interventions: Other: Dry needling; Other: Therapeutic Exercise
- Sham dry needling and exercise (Sham Comparator)
  Interventions: Other: Sham Dry Needling; Other: Therapeutic Exercise

INTERVENTIONS:
Other: Dry needling — Trigger point dry needling to trigger points in the shoulder or parascapular muscles using monofilament needle (i.e., acupuncture needle). Clean needle approach using sterile needles.
  Other Names: Trigger Point Dry Needling
  Arms: Dry needling and exercise
Other: Sham Dry Needling — Sham needle approach using a finishing nail in a tube sheath. The finishing nail will be placed over the trigger point so that the patient perceives a sharp sensation. The tube (not the nail) will be moved up and down to mimic the action of needling.
  Arms: Sham dry needling and exercise
Other: Therapeutic Exercise — Exercise including flexibility, range of motion, strengthening will be provided by the treating physical therapist based on the impairments identified.
  Other Names: Exercise

SUMMARY:
This study evaluates the addition of dry needling to exercise as part of physical therapy for the treatment of shoulder adhesive capsulitis. There will be two groups. One will receive actual dry needling to the clinically determined shoulder / parascapular trigger points. The other group will receive a sham needle treatment to the clinically determined areas.

DETAILED DESCRIPTION:
Shoulder adhesive capsulitis is reported to affect 2% to 5% of the general population. The clinical course of adhesive capsulitis has been described in the literature ranging from 18-24 months, with persistent symptoms often lasting longer after range of motion has returned. Fifty percent of individuals will report having mild pain or stiffness at 7-year follow up. Treatment for adhesive capsulitis can be extensive with the average duration of treatment being 4.7 months. In general, adhesive capsulitis is often thought of as a self limiting diagnosis that significantly impacts a patients function and livelihood. Physical therapists often prescribe exercise for the management of adhesive capsulitis including stretching and strengthening. There is some support for exercise to provide moderate improvements in function, mobility, and decreased pain but impairments including pain and range of motion deficits persist even with exercise treatments.

Trigger point dry needling is a treatment approach often used by physical therapists that has been purported to be effective for reducing pain and improving range of motion along with improving function. Improvements in range of motion are associated with improvements in function for patients with adhesive capsulitis. While dry needling does not directly treat the tissues thought to be the primary factor in limiting range of motion, it does treat the surrounding tissues, including trigger points, that have been associated with painful shoulders including adhesive capsulitis. However, the direct investigation of dry needling for shoulder adhesive capsulitis has been minimally investigated. While published papers on dry needling for adhesive capsulitis exists, they are primarily case reports or case series. The growth in utilization of dry needling as a treatment option with minimal evidence creates a dilemma in practice.

This will be a single blinded randomized controlled trial comparing dry needling with exercise versus sham dry needling and exercise for subjects with shoulder pain consistent with adhesive capsulitis.

Patients undergoing physical therapy examination for adhesive capsulitis will be considered for participation in the study. If the evaluating/treating physical therapist deems that the patient may be appropriate for the study, he/she will approach the patient to gauge interest in participating in the study. If the patient expresses interest, he or she will be referred to a member of the study personnel (dry needling physical therapist) who will screen for the inclusion and exclusion criteria. The study personnel will provide additional details regarding the study requirements. The consent process may be initiated at this time or deferred to a later time if the patient requests additional time to consider participation. After consenting, the patient will be randomly assigned to one of the two treatment groups. A digital coin flip (Siri) will be used for randomization procedures to determine the group allocation (dry needling and exercise or sham dry needling and exercise). Exercise prescription will be prescribed pragmatically. These will be based on the individual patient examination and re-examination findings by the treating physical therapists, and supported by best evidence. These exercises will address strength, flexibility and postural impairments based on the clinical examination. The treating physical therapist will be blinded to the dry needling treatment group assigned. The study personnel physical therapist will be blinded to the outcomes.

For subjects that are randomized to the group receiving trigger point dry needling, active and latent trigger points as described in previous protocols for dry needling of the shoulder will be used to determine the appropriate muscles to treat. The study personnel physical therapist will perform the dry needling (dry needling physical therapists). All dry needling physical therapists have had considerable and appropriate training in trigger point dry needling. Clean needle techniques will be applied including use of gloves by the physical therapist and chlorhexidine wipes (or alcohol wipes if a chlorhexidine allergy is known) for skin preparation. The dry needling procedure will involve using a sterile packaged Seirin ® 30-60 mm .25-.36 J-type monofilament needle. Palpation of the active or latent trigger point will direct the study personnel as to where to treat. The needle will be inserted using an insertion tube. Pistoning and twisting of the needle will be performed to elicit a local twitch response. The study personnel will document the muscle treated, if a local twitch response occurred, and if it was an active or latent trigger point. The frequency of dry needling sessions will be determined in part by the dry needling physical therapist as well as the subject. Subjects who defer subsuquent dry needling treatments will be noted accordingly in the database.

For subjects that are randomized to the group receiving sham dry needling group, the assessment procedure will be the same as the dry needling group. The same clean approach to needling will be performed in order to mimic the procedure of actual trigger point dry needling. Palpation of the active or latent trigger point will direct where to treat. The dry needling physical therapists will be trained by the principal investigator on the sham dry needling technique. A finishing nail cleaned with sterile alcohol swab will be inserted into a tube with the tip of the nail extended out the end of the tube. The physical therapist will use this sham needle over the area of the trigger point without skin penetration.

The finishing nail provides a minimal sharp sensation that is sometimes felt by patients receiving dry needling. It also matches the potential perception that a patient has regarding receiving any needle treatments. The force of the sham (finishing nail) treatment will be just enough to produce a slight sharp sensation. The tap provided is just enough so that the patient perceives a light sharp sensation. The procedure is set up similarly to actual dry needling in that the physical therapist uses the same finger and holding position of the tube. After the tap of the finishing nail, pseudo pistoning of the tube only (not the nail) will be performed to match the duration of treatment time of actual dry needling. This will range from 2 to 10 pistons varied per patient per muscle to match the approach of actual trigger point dry needling. Furthermore, the finishing nail will be held toward the base of the tube with firm pressure of the tube on the patient's skin to ensure consistent pressure is provided.

For both groups, the patient will be prone so that the patient remains blinded to the treatment. All set up procedures will take place after the patient has assumed the prone positon. After the patient has assumed the prone position, the treating physical therapist will prepare the treatment area as previously described. All materials associated with the intervention will be discarded and removed from the treatment area before the patient comes out of the prone position.

The duration of the total treatment program will be determined by the treating physical therapist based on the impairments and re-evaluation of the subjects status. Outcome measures will be collected at baseline. After one-month, or if the treating physical therapist deems the subject is appropriate for discharge (whichever comes first), all outcome measures will be reassessed. If the subject should need additional physical therapy after the one-month period, the physical therapist will document the types of interventions provided, and any additional healthcare utilization variables, including physical therapy utilization, and a final collection of outcomes. Follow up will be conducted at one-week, one-month (or discharge, whichever comes first) months and at 6 months to collect outcomes data.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of shoulder pain and stiffness
* Gradual onset of symptoms
* Glenohumeral passive range of motion limited in multiple directions
* Glenohumeral passive range of motion decreases as the humerus is abducted from 45 degrees to 90 degrees
* Age 18 to 65 years
* Reports pain with normal activity greater than or equal to 2/10 on the numeric pain rating scale
* Read and speak English

Exclusion Criteria:

* Signs or symptoms of cervical radiculopathy, radiculitis, or referral from the cervical spine
* Clinical evidence as determined in the examination of an alternative shoulder diagnosis
* Normal passive shoulder range of motion
* Known radiographic evidence of glenohumeral osteoarthritis
* Known neurologic disease
* Received dry needling or acupuncture within the past 6 months
* Fear of needling
* Currently being treated with anticoagulant medication
* Shoulder pain and disability index (SPADI) score less than 10% or greater than 90%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index Change | 1-week, 1-month, 6-months
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire. Two dimensions are measured, one for pain and the other for functional activities. The pain dimension includes five questions to determine the severity of an individual's pain. The functional activities are assessed with eight questions. The two dimensions are combined into one score. Scores range from 0 to 100 with scores closer to 0 indicating lower (or no) disability and scores closer to 100 indicating greater disability. It takes 5 to 10 minutes for a patient to complete.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale Change | 1-week, 1-month, 6- months
  The numeric pain rating scale (NPRS) is an 11 point scale scored between "0" (no pain) and "10" (the most intense pain imaginable). Individuals select a value that is most in the with the intensity of pain they've experienced in the past 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Clewley, DPT, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clewley D, Flynn TW, Koppenhaver S. Trigger point dry needling as an adjunct treatment for a patient with adhesive capsulitis of the shoulder. J Orthop Sports Phys Ther. 2014 Feb;44(2):92-101. doi: 10.2519/jospt.2014.4915. Epub 2013 Nov 21. PMID 24261931
- [Background] Dempsey AL, Mills T, Karsch RM, Branch TP. Maximizing total end range time is safe and effective for the conservative treatment of frozen shoulder patients. Am J Phys Med Rehabil. 2011 Sep;90(9):738-45. doi: 10.1097/PHM.0b013e318214ed0d. PMID 21430510
- [Background] Griggs SM, Ahn A, Green A. Idiopathic adhesive capsulitis. A prospective functional outcome study of nonoperative treatment. J Bone Joint Surg Am. 2000 Oct;82(10):1398-407. PMID 11057467
- [Background] Hall ML, Mackie AC, Ribeiro DC. Effects of dry needling trigger point therapy in the shoulder region on patients with upper extremity pain and dysfunction: a systematic review with meta-analysis. Physiotherapy. 2018 Jun;104(2):167-177. doi: 10.1016/j.physio.2017.08.001. Epub 2017 Aug 7. PMID 29439829
- [Background] Jewell DV, Riddle DL, Thacker LR. Interventions associated with an increased or decreased likelihood of pain reduction and improved function in patients with adhesive capsulitis: a retrospective cohort study. Phys Ther. 2009 May;89(5):419-29. doi: 10.2522/ptj.20080250. Epub 2009 Mar 6. PMID 19270045
- [Background] Koppenhaver S, Embry R, Ciccarello J, Waltrip J, Pike R, Walker M, Fernandez-de-Las-Penas C, Croy T, Flynn T. Effects of dry needling to the symptomatic versus control shoulder in patients with unilateral subacromial pain syndrome. Man Ther. 2016 Dec;26:62-69. doi: 10.1016/j.math.2016.07.009. Epub 2016 Jul 21. PMID 27497188
- [Background] Perez-Palomares S, Olivan-Blazquez B, Perez-Palomares A, Gaspar-Calvo E, Perez-Benito M, Lopez-Lapena E, de la Torre-Beldarrain ML, Magallon-Botaya R. Contribution of Dry Needling to Individualized Physical Therapy Treatment of Shoulder Pain: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2017 Jan;47(1):11-20. doi: 10.2519/jospt.2017.6698. Epub 2016 Dec 10. PMID 27937046
- [Background] Tejera-Falcon E, Toledo-Martel NDC, Sosa-Medina FM, Santana-Gonzalez F, Quintana-de la Fe MDP, Gallego-Izquierdo T, Pecos-Martin D. Dry needling in a manual physiotherapy and therapeutic exercise protocol for patients with chronic mechanical shoulder pain of unspecific origin: a protocol for a randomized control trial. BMC Musculoskelet Disord. 2017 Sep 18;18(1):400. doi: 10.1186/s12891-017-1746-3. PMID 28923050
- [Background] Sutlive TG, Golden A, King K, Morris WB, Morrison JE, Moore JH, Koppenhaver S. SHORT-TERM EFFECTS OF TRIGGER POINT DRY NEEDLING ON PAIN AND DISABILITY IN SUBJECTS WITH PATELLOFEMORAL PAIN SYNDROME. Int J Sports Phys Ther. 2018 Jun;13(3):462-473. PMID 30038832